CLINICAL TRIAL: NCT00013494
Title: Video-Based Functional Performance and Assessment Following Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: E2169T
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2006-03

CONDITIONS: Stroke
Keywords: Hemiplegia; elderly; Video; F-PAT,Functional Performance; digitized videoclips
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Stroke Rehabilitation

INTERVENTIONS:
Procedure: Stroke Rehabilitation

SUMMARY:
For hemiplegic, stroke patients wheelchair transfers is a critical, safety-related area of physical function.

This project will develop a personalized training and clinical assessment instrument based on the Video-Based F-PAT (Functional Performance Assessment and Training.) The objectives of the study are: (1) Enhance the pilot F-PAT web site to allow clinicians password-protected access to the digitized video and assessment information; and (2) train an Occupational Therapist collaborator to create the personalized videotapes for patients to take home with them. This study has the dual goal of evaluating the effectiveness of the personalized training videotapes and the effectiveness of the video-based assessment methodology.

DETAILED DESCRIPTION:
For people who have become hemiplegic as a result of a stroke, a critical safety-related retraining area for physical functions is wheelchair transfers. In addition, to incorporate the relatively unsupervised home care into the rehabilitation process, clinicians require a better means to assess functional gains and provide effective training tools. Our goal is to develop a personalized training and clinical assessment instrument based on the Video-Based F-PAT (Functional Performance Assessment and Training) which relies on the manipulation of digitized videoclips. Our development objectives are (1) to enhance the pilot F-PAT web site to allow clinicians password-protected access to the digitized video and assessment information; and (2) to train an Occupational Therapist collaborator to create the personalized videotapes for patients to take home with them. Our clinical objective is to implement a 2-year evaluation of the F-PAT design concept with 30 subjects, divided in 3 groups, who as patients undergo acute rehabilitation at the VA Comprehensive Rehabilitation Center and are discharged to their homes or a sub-acute facility. This study has the dual goal of evaluating the effectiveness of the personalized training videotapes and the effectiveness of the video-based assessment methodology.

The study will divide the subjects into three treatment groups to compare the effectiveness of accepted practice, generic videotape, and personalized videotape home-based instruction for clients and care providers. Comparison of outcomes will be done using videotape of task performance before release from the acute therapy program and at the follow-up evaluation one month later. The subjects will be evaluated by a blinded physiatrist viewing and rating digitized videoclips of task performance on the F-PAT web site. This study will determine if personalized videoclip-based instructional material is effective, and if videoclip comparisons by a clinician is an effective diagnosis and assessment instrument. If it is not possible for logistical reasons for a subject to return to the clinic for the follow-on evaluation, the F-PAT team will visit the subject's home and perform the videotaping on-site. The remainder of the evaluation with input from the physiatrist will occur subsequently at the clinic.

ELIGIBILITY:
Hemiplegic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 1999-07; Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fryer, Ph.D., Asst. Director — Department of Veterans Affairs, Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service; Victoria Mongiardo, Program Analyst — Department of Veterans Affairs, Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service
Locations (1):
- VAMC, Palo Alto, Palo Alto, California, United States